CLINICAL TRIAL: NCT04752254
Title: Cognitive Hyperarousal in Insomnia Disorder
Brief Title: Investigating Racing Thoughts in Patients With Insomnia Disorder
Acronym: TIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7987
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Hyperarousal; Rumination; Racing thoughts
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Rumination Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cognitive arousal has been identified as playing a key role in the inability to fall asleep or stay asleep. However, although people with insomnia frequently complain about racing thoughts appearing as soon as they get into bed, studies focusing on racing thoughts in insomnia are lacking. The aim of the present study is to investigate racing thoughts in insomnia disorder using a self-report questionnaire, the Racing and Crowded Thoughts Questionnaire. Specifically, the researchers seek to address three related goals: the comparison of RCTQ scores in adults with primary insomnia, healthy individuals, and patients with bipolar disorder in a manic/hypomanic episode; the variation of RCTQ scores relative to time of day; and the specific contribution of racing thoughts to insomnia severity, as compared to worry and rumination.

ELIGIBILITY:
Inclusion Criteria:

* Major subject from 18 to 70 years old)
* with a diagnosis of chronic primary insomnia according to the criteria of ICSD-3
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice
* Patient with secondary insomnia (OSA, circadian rhythm disorder, severe restless legs syndrome, bipolar disorder, ADD +/- H)
* Subject under psychotropic treatment other than hypnotics
* Incomplete data concerning the main endpoint

Ages: 18 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with a diagnosis of chronic primary insomnia according to the criteria of ICSD-3
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
A retrospective evaluation of self-reported tachypsychia in primary insomnia | Files analysed retrospectively from Jun 01, 2014 to March 13, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sleep Disorders - CIRCSom - Strasbourg University Hospitals, Strasbourg, France

REFERENCES:
- [Derived] Weiner L, Martz E, Kilic-Huck U, Siegel N, Bertschy G, Geoffroy PA, Weibel S, Bourgin P. Investigating racing thoughts in insomnia: A neglected piece of the mood-sleep puzzle? Compr Psychiatry. 2021 Nov;111:152271. doi: 10.1016/j.comppsych.2021.152271. Epub 2021 Sep 17. PMID 34555554